CLINICAL TRIAL: NCT07208006
Title: Impact of PCSK9 Monoclonal Antibody Very Early Administered in Hospital to Reduce Cardiovascular Events in Acute Myocardial Infarction (IMMEDIATE -MI)
Brief Title: Very Early PCSK9 Inhibition for Acute Myocardial Infarction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2025169
Record Dates: First submitted 2025-09-27; First posted 2025-10-06 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-09

CONDITIONS: Acute Myocardial Infarction (AMI)
Keywords: Acute Myocardial Infarction; Multivessel Disease; PCSK9 Inhibitor; Lipid-Lowering Therapy; Plaque Vulnerability; MACE

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Lipid-Lowering Therapy (Active Comparator): Participants will receive guideline-recommended lipid-lowering therapy starting with statins. Based on follow-up lipid levels, additional agents such as ezetimibe and PCSK9 inhibitors may be added sequentially, according to routine clinical practice.
  Interventions: Drug: Standard Lipid-Lowering Therapy
- Early Intensive Lipid-Lowering Therapy (PCSK9 Inhibitor) (Experimental): Participants will receive early intensive lipid-lowering therapy with a PCSK9 monoclonal antibody initiated during index hospitalization, in addition to statins. Ezetimibe may be added as needed. The PCSK9 inhibitor will be given regardless of baseline lipid levels.
  Interventions: Drug: Early Intensive Lipid-Lowering Therapy (PCSK9 Inhibitor)

INTERVENTIONS:
Drug: Standard Lipid-Lowering Therapy — Participants will receive lipid-lowering therapy according to current clinical guidelines. Treatment will be initiated with statins. Based on follow-up lipid levels, ezetimibe may be added, and PCSK9 inhibitor therapy may be considered if LDL-C goals are not met.
  Arms: Standard Lipid-Lowering Therapy
Drug: Early Intensive Lipid-Lowering Therapy (PCSK9 Inhibitor) — Participants will receive early intensive lipid-lowering therapy with a PCSK9 monoclonal antibody, initiated during the index hospitalization, in addition to statins. Ezetimibe may be added if clinically indicated. The PCSK9 inhibitor will be administered regardless of baseline lipid levels.
  Arms: Early Intensive Lipid-Lowering Therapy (PCSK9 Inhibitor)

SUMMARY:
Acute myocardial infarction (AMI) remains a major cause of morbidity and mortality, particularly in patients with multivessel coronary artery disease. Although primary percutaneous coronary intervention (PCI) has significantly improved short-term outcomes, these patients remain at high risk of recurrent cardiovascular events due to vulnerable non-culprit plaques. Coronary imaging techniques such as intravascular ultrasound (IVUS), optical coherence tomography (OCT), and angiography-derived indices (QFR, RWS) can identify high-risk lesions, but the optimal management strategy is still debated.

Early and intensive lipid-lowering therapy has been shown to stabilize atherosclerotic plaques. PCSK9 monoclonal antibodies, in combination with statins, provide rapid and profound LDL-cholesterol reduction and may enhance plaque stabilization beyond standard therapy. Small imaging studies suggest favorable effects of PCSK9 inhibitors on fibrous cap thickness and lipid burden, but their impact on clinical outcomes in AMI patients with multivessel disease remains uncertain.

This study aims to evaluate whether very early in-hospital administration of a PCSK9 inhibitor, in addition to standard care, can reduce major adverse cardiovascular events (MACE) over 12 months compared with standard lipid-lowering therapy alone. The trial will also explore imaging-based markers of plaque vulnerability and functional indices as secondary endpoints, in order to better understand the mechanisms linking lipid lowering, plaque stabilization, and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥18 years.
2. Acute myocardial infarction (AMI) onset within 30 days (first hospitalization with a confirmed diagnosis of STEMI or NSTEMI).
3. Multivessel coronary artery disease; successful percutaneous coronary intervention (PCI) of the culprit lesion in the infarct-related artery (IRA), including stent implantation and/or balloon angioplasty and/or thrombus aspiration.
4. At least one angiographically assessed diameter stenosis ≥50% in a non-infarct-related artery (non-IRA) with a reference vessel diameter ≥2.5 mm.
5. Able to understand and willing to provide written informed consent, comply with prescribed medical therapy, and complete the required follow-up.

Exclusion Criteria

1. Cardiogenic shock or severe heart failure (Killip class IV).
2. Serum creatinine >150 μmol/L or glomerular filtration rate (GFR) <45 mL/min/1.73 m² calculated by the Cockcroft-Gault equation.
3. Known or suspected infective endocarditis or active systemic infection.
4. Clinically significant coagulation abnormalities, or anticipated inability to tolerate long-term antiplatelet therapy.
5. Pregnant or breastfeeding women, women planning pregnancy within 1 year, or those unwilling to use effective contraception.
6. Expected survival <1 year.
7. Allergy to iodinated contrast media.
8. Prior coronary artery bypass grafting (CABG).
9. Participation in another clinical trial within 3 months before enrollment, or current participation in another drug/device clinical trial without having reached its primary endpoint.
10. Coronary angiography-based exclusion criteria:

10.1 Non-IRA lesion with visually estimated diameter stenosis >90% and TIMI flow ≤2; 10.2 Complex coronary artery disease requiring CABG; 10.3 Angiography unable to clearly identify the infarct-related artery or non-infarct-related arteries.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1518 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Major Adverse Cardiovascular Events (MACE) at 12 Months | 12 months after index percutaneous coronary intervention (±30 days)
  MACE is defined as a composite endpoint including all-cause death, non-fatal myocardial infarction, stroke, unplanned ischemia-driven revascularization, and rehospitalization for unstable angina. The occurrence of the first event from this composite will be recorded for each participant.

SECONDARY OUTCOMES:
Incidence of Key Secondary Cardiovascular Events | 12 months after index PCI (±30 days)
  Composite of cardiovascular death, non-fatal myocardial infarction, stroke, and unplanned ischemia-driven revascularization.
Incidence of All-Cause Death | 12 months after index PCI (±30 days)
  Death from cardiovascular causes, non-cardiovascular causes, or unknown causes.
Incidence of Non-fatal Myocardial Infarction | 12 months after index PCI (±30 days)
  Defined according to SCAI criteria for peri-procedural MI and spontaneous MI related to culprit or non-culprit vessels.
Incidence of Non-fatal Ischemic Stroke | 12 months after index PCI (±30 days)
  Stroke confirmed by clinical diagnosis and imaging, excluding hemorrhagic stroke.
Incidence of Unplanned Ischemia-Driven Revascularization | 12 months after index PCI (±30 days)
  Repeat PCI or CABG driven by ischemic symptoms or objective evidence of ischemia, involving culprit or non-culprit vessels.
Rehospitalization for Unstable Angina | 12 months after index PCI (±30 days)
  Hospital admission due to recurrent chest pain confirmed as unstable angina requiring medical management.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No